CLINICAL TRIAL: NCT06033378
Title: Blood Pressure Treatment in ICU Patients with Subarachniodal Haemorrhage. -Can Blood Pressure Be Used As a Surrogate Marker for Blood Flow
Brief Title: Blood Pressure Treatment in ICU Patients with Subarachniodal Haemorrhage.
Acronym: BFBP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Region Västerbotten (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2022-06754-01
Record Dates: First submitted 2023-09-04; First posted 2023-09-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-02

CONDITIONS: Blood Pressure; Subarachnoid Hemorrhage; Aneurysm Cerebral
Keywords: magnetic resonance imaging; norepinephrine; blood flow
MeSH Terms: conditions — Subarachnoid Hemorrhage; Intracranial Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cerebral blood flow (Experimental): Change in cerebral blood flow with increased systemic blood pressure
  Interventions: Other: Blood pressure elevation

INTERVENTIONS:
Other: Blood pressure elevation — Increasing systemic blood pressure for measurement of cerebral blood flow changes

SUMMARY:
An MRI study to examine the relationship between blood pressure and cerebral blood flow in patients with subarachnoidal hemorrhage and suspect or verified vasospasm.

DETAILED DESCRIPTION:
Subarachnoidal hemorrhage (SAH) is a type of stroke with high mortality rates and often requires care at the intensive care unit. Cerebral blood flow (CBF) needs to be ensured so that the brain receives optimal nourishment, and this is largely controlled by regulating blood pressure (BP) using medications that affect the heart and blood vessels. Approximately 3-7 days after SAH onset, vasospasm (SAH-V) can occur. Treatment usually includes maintaining blood pressure (BP) above a certain threshold to achieve adequate cerebral blood flow (CBF). An important component of raising BP is increasing vascular resistance using vasoconstrictive medications, which paradoxically can decrease CBF.

The study objective is to investigate the correlation between BP changes and their impact on CBF in patients with suspect or verified SAH-V using MRI.

To achieve this purpose, the investigators plan to examine the relationship between BP and CBF in patients with SAH-V who require neuro-intensive care. To measure CBF, two techniquis will be used: phase-contrast MRI and arterial spin labeling.

Flow measurement with MRI:

1. Baseline images will be acquired at baseline blood pressure.
2. Mean arterial pressure (MAP) will be increased using norepinephrine. New images will be acquired when MAP is increased by approximately 20-30% from the baseline.

All BP levels will be maintained within clinically acceptable ranges. All data will be recorded in the patient's medical record, and MRI images will be processed at a later stage.

ELIGIBILITY:
Inclusion Criteria:

* Coiled or clipped aneurysm
* Suspected or confirmed vasospasm

Exclusion Criteria:

* BMI >30
* Pregnancy
* Pacemaker or other MRI contraindications
* Severe congestive heart failure (NYHA III-IV) or cardiac arrhythmia.
* Severe respiratory failure or FiO2 >0.6
* Severe kidney failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Cerebral blood flow | 1 hour
  mL/min as measured by MRI

CONTACTS AND LOCATIONS:
Overall Officials: Laleh Zarrinkoob, Principal Investigator — Region Västerbotten
Locations (1):
- Umeå University Hospital, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Osterlind J, Birnefeld J, Birnefeld E, Hultin M, Qvarlander S, Wahlin A, Holmlund P, Zarrinkoob L. Study protocol: MRI-based assessment of cerebral blood flow under pharmacologically elevated blood pressure in patients under general anesthesia, and in sedated ICU patients with aneurysmal subarachnoid hemorrhage. PLoS One. 2025 Dec 10;20(12):e0338688. doi: 10.1371/journal.pone.0338688. eCollection 2025. PMID 41370289